CLINICAL TRIAL: NCT05458180
Title: Phase I Cinical Sudy of Lposomal Mitoxantrone Hydrochloride Combined With Cyclophosphamide, Vincristine, Etoposide and Prednisone (CMOEP) in Previously Untreated Peripheral T-cell Lymphoma
Brief Title: CMOEP in the Treatment of Untreated Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-PTCL-K02
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMOEP (Experimental): dose-escalation： Untreated Peripheral T-cell Lymphoma Patients will receive sequentially higher doses of liposomal mitoxantrone hydrochloride in combination with Cyclophosphamide, Vincristine, Etoposide and Prednisone for 6 cycles (planned) (21 days per cycle). The initial dose of liposomal mitoxantrone hydrochloride is 15 mg/m2.
  Interventions: Drug: Lposomal mitoxantrone hydrochloride,Cyclophosphamide,Vincristine,Etoposide and Prednisone(CMOEP)

INTERVENTIONS:
Drug: Lposomal mitoxantrone hydrochloride,Cyclophosphamide,Vincristine,Etoposide and Prednisone(CMOEP) — Drug: Liposomal mitoxantrone hydrochloride (15 mg/m2, 18 mg/m2, 20 mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Drug: Cyclophosphamide (750 mg/ m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Drug: Vincristine (1.4mg/ m2，Max dose 2mg) will be administered by an intravenous injection on day 1of each 21-day cycle.
  Drug: Etoposide (60 mg/ m2) will be administered by an intravenous infusion on day 1-3 of each 21-day cycle.
  Drug: Prednisone (100 mg) will be taken orally from day 1-5 of each 21-day cycle.

SUMMARY:
This is a prospective, single arm, multicenter, dose-escalation clinical study to evaluate the safety and efficacy of CMOEP in patients with untreated Peripheral T-cell Lymphoma.

DETAILED DESCRIPTION:
This is a single arm, multicenter, dose-escalation study which mainly explores the dose limiting toxicity (DLT) of liposomal mitoxantrone hydrochloride in combination with Cyclophosphamide, Vincristine, Etoposide and Prednisone（CMOEP） in patients with untreated Peripheral T-cell Lymphoma. Liposomal mitoxantrone hydrochloride will be given on day 1 at three different doses (15 mg/m2, 18 mg/m2, 20 mg/m2) and be combined with Cyclophosphamide, Vincristine, Etoposide and Prednisone. The dose limited toxicity (DLT) will be evaluated after the first cycle of therapy. A maximum of 6 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent.
2. Age ≥18, ≤65years, no gender limitation.
3. Expected survival ≥ 3 months.
4. Histologically confirmed diagnosis of Peripheral T-cell lymphoma： 1) Peripheral T-cell lymphoma unspecified (ptcl-NOS) 2) Angioimmunoblastic T-cell lymphoma (AITL) 3) Anaplastic large T-cell lymphoma (ALCL), ALK+ 4) Anaplastic large T-cell lymphoma (ALCL), ALK- 5) Other subtypes of PTCL that the investigator think can be included in the group.
5. No previous treatment for PTCL, including chemotherapy, targeted therapy, immunotherapy, local radiotherapy for lymphoma (except for local radiotherapy to alleviate tumor related symptoms), surgical treatment.
6. Subjects must have at least one evaluable or measurable lesion per lugano2014 criteria: for lymph node lesions, the length and diameter should be > 1.5cm; For non-lymph node lesions, the length and diameter should be > 1.0cm.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
8. The following baseline laboratory criteria are required: Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count (PLT) ≥75×10^9/L, Hemoglobin(HB)≥ 90 g/L.
9. Total Serum creatinine (Scr) ≤1.5X upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5X ULN, bilirubin (TBIL)≤1.5X ULN.

Exclusion Criteria:

1. The subject had previously received any of the following anti-tumor treatments:1）Subjects who have been treated with mitoxantrone or mitoxantrone liposomes;2）Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin was more than 360 mg/m2 (1 mg doxorubicin equivalent to 2 mg epirubicin).
2. Hypersensitivity to any study drug or its components.
3. Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.)
4. Heart function and disease meet one of the following conditions:1）Long QTc syndrome or QTc interval > 480 ms;2）Complete left bundle branch block, grade II or III atrioventricular block;3）Serious and uncontrolled arrhythmias requiring drug treatment;4）New York Heart Association grade ≥ II;5）Cardiac ejection fraction (LVEF)< 50%;6）A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
5. Hepatitis B and hepatitis C active infection (defined as hepatitis B virus surface antigen positive and hepatitis B virus DNA higher than 1x10^3 copy/mL; hepatitis C virus RNA high than 1x10^3 copy/mL).
6. Human immunodeficiency virus (HIV) infection (HIV antibody positive).
7. Patients with other malignant tumors, except for effectively controlled non melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ and other tumor during the past 5 years.
8. Patients with primary or secondary central nervous system (CNS) lymphoma or history of CNS lymphoma.
9. Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures.
10. Unsuitable subjects for this study determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-07-07 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Cycle 1 (21 days)
  Maximum tolerated dose (MTD) of liposomal mitoxantrone hydrochloride in CMOEP

SECONDARY OUTCOMES:
Dose limited toxicities (DLTs) | Cycle 1 (21 days)
  Adverse events (AE) defined as DLT events per protocol
The incidence of AE and SAE | Up to 28 days after the last patient complete his study therapy
  AE or severe adverse events (SAE) occur since the first dose of therapy is given
Objective response rate (ORR) | Up to 1 year
  Response is assessed according to the lugano criteria
Complete response rate (CRR) | Up to 1 year
  Response is assessed according to the lugano criteria
Progression-free survival（PFS） | Up to 1 year
  From the date of the first dose of therapy is given until disease progression, death

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared with other researchers

REFERENCES:
- [Derived] Yu J, Sun X, Gao G, Yu L, Wang J, Qiu L, Qian Z, Li W, Zhang H. CMOEP regimen in the treatment of untreated peripheral T-cell lymphoma: a multicenter, single-arm, phase I study. Front Immunol. 2025 Apr 11;16:1551723. doi: 10.3389/fimmu.2025.1551723. eCollection 2025. PMID 40292284